CLINICAL TRIAL: NCT00418587
Title: Phase 1 Study of Vitamin D Therapy in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Vitamin D Therapy in Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American College of Rheumatology Research and Education Foundation (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUSC-GAC734-HR16356
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Vitamin D; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 800 IU oral daily dose level
  Interventions: Drug: Cholecalciferol
- 2 (Experimental): 2000 IU oral daily dose level
  Interventions: Drug: Cholecalciferol
- 3 (Experimental): 4000 IU oral daily dose level
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 800 IU oral daily
  Other Names: Vitamin D3
  Arms: 1
Drug: Cholecalciferol — 2000 IU oral daily
  Other Names: Vitamin D3
  Arms: 2
Drug: Cholecalciferol — 4000 IU oral daily
  Other Names: Vitamin D3
  Arms: 3

SUMMARY:
The purpose of this study is to test the safety and effectiveness of different doses of vitamin D in patients with Systemic Lupus Erythematosus (SLE). A long term goal is to determine if vitamin D could be used as a treatment and/or preventative of SLE.

ELIGIBILITY:
Inclusion Criteria:

* SLE by ACR criteria (revised 1997)
* African American, participating in the SLE in Gullah Health (SLEIGH) Study
* Outpatient
* Stable disease with no BILAG A or B in any system for the past 4 weeks
* Stable prednisone (or equivalent corticosteroid) dose ≤ 20 mg/day for ≥ 4 weeks prior to study entry
* Baseline 25(OH)D concentration of < 30 ng/ml
* Willingness to discontinue other vitamin D supplements and/or multivitamins containing vitamin D while participating in the study
* Age 18 - 85 years
* Ability to complete questionnaires in English
* Ability to give informed consent

Exclusion Criteria:

* Presence of hypercalcemia (>10.4 mg/dL), hypercalcuria (urinary calcium/creatinine ratio ≥ 0.8 mmol/mmol) or known primary hyperparathyroidism
* Liver disease (serum ALT, AST >2x normal) or total serum bilirubin >1.5x normal
* History of renal stones
* Current treatment with any dose of cyclophosphamide
* Dialysis or creatinine > 2.5 mg/dL
* Pregnancy
* Current drug or alcohol abuse
* Anticipated poor compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hypercalcuria | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Kamen, MD, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States